CLINICAL TRIAL: NCT03388697
Title: Validation of a Novel Screening Test for Maternal Insulin Resistance and Predicting Maternal Fetal Outcomes: A Pilot Study.
Brief Title: Validation of a Novel Screening Test for Maternal Insulin Resistance
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 17-0228
Record Dates: First submitted 2017-12-07; First posted 2018-01-03 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2019-02

CONDITIONS: Insulin Resistance, Diabetes
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Two tubes (total = 20cc) of blood will be collected from participants who will be asked to fast for minimum of 8 hours prior to blood draw.
  The samples from both time points will be sent together to Metabolon for Quantose IR and Quantose IGT analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Quantose IR and Quantose IGT analysis — Testing using Quantose IR and Quantose IGT: The blood draws will be timed to coincide with clinically indicated blood tests as much as possible (e.g. first visit labs, aneuploidy screening, gestational diabetes screening).
  Other Names: QUANTOSE® IR, QUANTOSE® IGTT
Diagnostic Test: HOMA IR the standard testing for insulin resistance — Testing using HOMA IR: Investigators will be measuring fasting insulin and glucose levels (last meal more than 8hrs before testing i.e. overnight fasting) from EDTA-plasma samples. After collection, the samples will be spun and plasma obtained. Samples will be stored until testing. The investigators will be using the following computation to calculate HOMA.
  Other Names: HOMA IR

SUMMARY:
This will be a validation study of Quantose IR and Quantose IGT to predict insulin resistance and identify patients with prediabetes. This is a pilot study of 100 subjects. Based on the results of this initial trial, investigators plan to perform a larger trial at UTMB.

Quantose IR is a fasting blood test for insulin resistance and prediabetes, and is clinically validated in non-pregnant individuals. The Quantose IR Score is based on three novel nonglycemic biomarkers, as well as insulin, and provides a comprehensive measure of insulin resistance. These analytes include:

* α-HB (α-hydroxybutyrate): positively correlated with insulin resistance and indicative of early β-cell dysfunction.
* L-GPC (linoleoyl-glycerophosphocholine): negatively correlated with insulin resistance and impaired glucose tolerance.
* Oleic Acid: positively correlated with increasing lipolysis and insulin resistance.
* Insulin: increased insulin is characteristic of insulin resistance and is an independent risk factor for type 2 diabetes and cardiovascular disease.

Quantose IGT is designed to estimate the risk of being IGT. It is calculated from a multiple logistic regression model based on the fasting plasma levels of:

* Glucose.
* α-HB.
* β-HB.
* 4-methyl-2-oxopentanoic acid.
* LGPC.
* Oleic acid.
* Serine.
* Vitamin B5. Participants in the study will be consenting to data collection and two visits for lab draw. The investigators will then evaluate the performance of the Quantose IR and Quantose IGT in the study population.

DETAILED DESCRIPTION:
This is a prospective cohort non-interventional study. Subjects will be identified during the time of a prenatal visit at one of the UTMB clinics. All necessary institutional and regulatory approval will be obtained prior to enrolling any candidates for this study.

Potential subjects that are not patients of the investigator or patients of the study team members, they will not be contacted by study staff unless they have been informed of the study by their medical provider and express an interest in receiving more information on the study or wish to enroll in the study. Under the direction of the PI, trained research staff will be available in the UTMB prenatal care clinics to screen and consent subjects according to study protocol. The Perinatal Research Division (PRD) has staff based in the UTMB Maternal Health (OB) clinics. These research staff members will screen the charts and electronic medical records of prenatal patients receiving care in the OB clinics. In order to contact potential study participants, the HIPAA waiver is submitted.

In addition, the OB clinic staff will be in serviced on the study and encouraged to refer potential subjects to the PRD staff. Other than the blood samples for this study, the management of pregnancy and delivery will be according to the standard of care at UTMB and will be up to the clinical provider.

Blood samples will be collected during 2 windows, early window (gestational age 10 0/7 to 13 6/7 weeks) and late window (gestational age 24 0/7 to 28 0/7 weeks) and stored at -800C in our perinatal research division. An aliquot will be sent to Metabolon to run the Quantose IR and Quantose IGT. The laboratory and the investigators will be blinded to the outcomes of the patient.

Testing using Quantose IR and Quantose IGT: The blood draws will be timed to coincide with clinically indicated blood tests as much as possible (e.g. first visit labs, aneuploidy screening, gestational diabetes screening).

Testing using HOMA IR: The investigators will be measuring fasting insulin and glucose levels (last meal more than 8hrs before testing i.e. overnight fasting) from EDTA-plasma samples. After collection, the samples will be spun and plasma obtained. Samples will be stored until testing.

Two tubes (total = 20cc) of blood will be collected from participants who will be asked to fast for minimum of 8 hours prior to blood draw.

The samples from both time points will be sent together to Metabolon for Quantose IR and Quantose IGT analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Singleton pregnancy.
* Able to provide consent.
* Gestational age 10 0/7 to 13 6/7 weeks.
* Planned delivery at UTMB (John Sealy Hospital (JSH) or League City Hospital Campus.
* Pre-pregnancy or early pregnancy BMI > or = 30 kg/m2

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: * Known or suspected fetal anomaly.
  * Pre-gestational diabetes.
  * Pre-pregnancy hypertension.
  * Receiving medication that would interfere with Quantose IR or would increase IR (e.g. steroids).
  * Prisoners.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Gestational Diabetes | Up to 28 0/7 weeks of gestation
  Development of gestational diabetes (based on the two step approach: 1hr glucose screen > 135mg/dL and 2/4 abnormal values in a 3 hr OGTT using the Carpenter and Coustan

SECONDARY OUTCOMES:
Insulin resistance | Up to 28 0/7 weeks of gestation
  Defined as abnormal HOMA IR
Fasting Plasma glucose | Up to 28 0/7 weeks of gestation
  Measuring plasma glucose
Fasting Insulin | Up to 28 0/7 weeks of gestation
  Measuring plasma insulin level
1 hour glucola | Up to 28 0/7 weeks of gestation
  after receiving 50grams glucose load po and plasma glucose level is drawn 1 hour later
Perinatal death | up to 7 days after delivery
  stillbirths plus early neonatal deaths (under 7 days)
Neonatal hypoglycemia | up to 7 days after delivery
  Neonate plasma glucose < 90mg/dL
NICU admission | up to 7 days after delivery
  Admission to the neonatal intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Saad, MD, Principal Investigator — UTMB Galveston
Locations (1):
- Ashley Salazar, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ginsberg H, Olefsky JM, Reaven GM. Further evidence that insulin resistance exists in patients with chemical diabetes. Diabetes. 1974 Aug;23(8):674-8. doi: 10.2337/diab.23.8.674. No abstract available. PMID 4852112
- [Background] Harris MI. Epidemiologic studies on the pathogenesis of non-insulin-dependent diabetes mellitus (NIDDM). Clin Invest Med. 1995 Aug;18(4):231-9. PMID 8549007
- [Background] Lyssenko V, Jonsson A, Almgren P, Pulizzi N, Isomaa B, Tuomi T, Berglund G, Altshuler D, Nilsson P, Groop L. Clinical risk factors, DNA variants, and the development of type 2 diabetes. N Engl J Med. 2008 Nov 20;359(21):2220-32. doi: 10.1056/NEJMoa0801869. PMID 19020324
- [Background] Reaven GM. Insulin resistance and human disease: a short history. J Basic Clin Physiol Pharmacol. 1998;9(2-4):387-406. doi: 10.1515/jbcpp.1998.9.2-4.387. PMID 10212844
- [Derived] Eid J, Kechichian T, Benavides E, Thibodeaux L, Salazar AE, Saade GR, Saad AF. The Quantose Insulin Resistance Test for Maternal Insulin Resistance: A Pilot Study. Am J Perinatol. 2022 Apr;39(5):513-518. doi: 10.1055/s-0040-1716730. Epub 2020 Sep 7. PMID 32894869